CLINICAL TRIAL: NCT00458367
Title: Risperdal Safety Protocol Evaluation Consta Treatment; A Post Authorization Safety Survey With RISPERDAL CONSTA TM
Brief Title: RiSPECT: Risperdal Safety Protocol Evaluation Consta Treatment, a Post Authorization Safety Survey to Obtain Information on the Safety and Efficacy of Risperidone When Used in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: European Medical Affairs Director, Psychiatry, Janssen-Cilag S.A., Spain
Other Study IDs: CR003373
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Schizophrenia; Psychotic Disorders; Schizoaffective Disorder
Keywords: PASS; Safety Assessment; Efficacy Assessment; long-acting injectable risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: Open label risperidone long acting injectable intramuscular injections every 2 weeks for 26 weeks flexible dose 25 to 50 mg
  Interventions: Drug: Open label risperidone long acting injectable

INTERVENTIONS:
Drug: Open label risperidone long acting injectable — intramuscular injections every 2 weeks for 26 weeks, flexible dose 25 to 50 mg

SUMMARY:
The purpose of this research study is to gather information on the safety and efficacy of risperidone when used in routine clinical practice.

DETAILED DESCRIPTION:
This post-authorisation safety survey (PASS) is an international, multicentre, naturalistic, descriptive survey to confirm safety of risperidone in daily practice. This is a single-arm, prospective, observational survey to compare the safety profile between groups defined by existing risk or disease factors or patient characteristics. The study duration is 6 months with 4 patient visits. The primary objective of this PASS is to confirm safety, as identified in phase III clinical trials of risperidone, by collecting data when the drug is used under marketed conditions in routine clinical practice. A secondary objective is to evaluate effectiveness and reasons for initiating risperidone. Each investigator is to document data for 4-10 treated patients for whom risperidone long-acting injectable (RLAI) treatment is determined to be clinically indicated. Risperidone long-acting injectable (RLAI) is given as intramuscular injections every 2 weeks. The starting dose of RLAI will be in accordance with the product label (usually 25 mg). If necessary, the dosage of the injection may be increased gradually. Treatment duration is 26 weeks. To ensure continued antipsychotic coverage until the main release of risperidone from the microspheres, previous antipsychotic therapy will be continued concomitantly during the first three weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with long-acting injectable risperidone as decided after agreement between the physician and the patient, in accordance with the local Summary of Product Characteristics (SmPC), are eligible for inclusion in this survey. According to the global SmPC, long-acting injectable risperidone is indicated for the treatment of schizophrenia and schizoaffective disorder

Exclusion Criteria:

* According to the SmPC, long-acting injectable risperidone is contraindicated in patients with a known hypersensitivity to the product or any of its components. These patients must be excluded from the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with long-acting injectable risperidone as decided after agreement between the physician and the patient, in accordance with the local SmPC, are eligible for inclusion in this survey. According to the global SmPC, long-acting injectable risperidone is indicated for the treatment of schizophrenia and schizoaffective disorder.
Sampling Method: Non-Probability Sample
Enrollment: 5296 (Actual)
Dates: Start 2002-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To confirm safety, as identified in phase III clinical trials of risperidone by collecting data (including adverse event information) when the drug is used under marketed conditions in routine clinical practice. | at baseline and at month 1, 3 and 6.

SECONDARY OUTCOMES:
To evaluate effectiveness of risperidone long acting injectable (using Clinical Global Impression scale-Severity and Change) | Baseline and at month 1, 3 and 6
To evaluate effectiveness of risperidone long acting injectable (using Global Assessment of Functioning scale) | Baseline and at month 1, 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.